CLINICAL TRIAL: NCT04152941
Title: Observational Retrospective Cohort Study in Patients With Relapsed Epithelial Ovarian, Fallopian Tube, or Peritoneal Cancer Treated With Olaparib Following Response to Platinium-based Chemotherapy
Brief Title: Real-life Data of Olaparib in Relapsed Ovarian Cancers Patients
Acronym: RETROLA
Status: Completed | Type: Observational
Sponsor: ARCAGY/ GINECO GROUP (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: GINECO-OV-237
Record Dates: First submitted 2019-10-22; First posted 2019-11-06 (Actual); Last update posted 2023-09-06 (Actual); Status verified 2023-09

CONDITIONS: Relapsed Ovarian Cancers Patients
MeSH Terms: interventions — olaparib

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Olaparib — Patients with histologically confirmed ovarian cancer, primary peritoneal cancer and / or fallopian-tube cancer treated with olaparib in a real life-setting, between May 2014 to March 2017, whatever the line of therapy

SUMMARY:
This is a national, multi center, retrospective observational cohort study that will be carried out by reviewing the medical records of patients with relapsed epithelial ovarian, fallopian tube, or peritoneal cancer treated with olaparib following response to platinum-based chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be female ≥18 years of age
* Patients with histologically confirmed ovarian cancer, primary peritoneal cancer and / or fallopian-tube cancer that were treated with olaparib in a real life-setting, between May 2014 to March 2017, whatever the line of therapy
* Patients can be either alive or deceased at the time of medical record abstraction
* Patients should not have any objection that anonymized data will be collected and subjected to automated processing.

Exclusion Criteria:

* Patient that were given olaparib within a clinical trial

Min Age: 18 Years | Sex: Female
Age Groups: Adult, Older Adult
Study Population: The patient population observed in this study must fulfil all of the following inclusion criteria:
  * Patients must be female ≥18 years of age
  * Patients with histologically confirmed ovarian cancer, primary peritoneal cancer and / or fallopian-tube cancer that were treated with olaparib in a real life-setting, between May 2014 to March 2017, whatever the line of therapy
  * Patients can be either alive or deceased at the time of medical record abstraction
  * Patients should not have any objection that anonymized data will be collected and subjected to automated processing.
Sampling Method: Non-Probability Sample
Enrollment: 130 (Actual)
Dates: Start 2018-10-11 (Actual); Primary Completion 2020-02-11 (Actual); Study Completion 2020-02-11 (Actual)

PRIMARY OUTCOMES:
progression free survival (PFS) | through study completion, an average of 1 year
  PFS (days) = date of progression - date of treatment start + 1
overall Survival (OS) | through study completion, an average of 1 year
  OS (days) = date of death - date of treatment start + 1
incidence of events of clinical interest | through study completion, an average of 1 year
  the following events: anemia, thrombopenia, nausea and vomiting, fatigue, myelodysplastic syndrome, upper respiratory infections, diarrhea, decreased appetite, dysgeusia and headache will be formally retrieved from the source documents.

CONTACTS AND LOCATIONS:
Overall Officials: Thibault de La Motte Rouge, Dr, Principal Investigator — Centre Eugène Marquis
Locations (28):
- France (28):
  - ICO Paul Papin, Angers
  - Institut Sainte-Catherine, Avignon
  - CHRU Jean Minjoz, Besançon
  - Clinique Tivoli, Bordeaux
  - Institut Bergonié, Bordeaux
  - Clinique Pasteur, Brest
  - Hôpital Morvan - Centre Hospitalier Universitaire, Brest
  - Centre Jean Perrin, Clermont-Ferrand
  - Centre Georges François Leclerc, Dijon
  - Groupe Hospitalier Mutualiste de Grenoble, Grenoble
  - Institut Hospitalier Franco-Britannique, Levallois-Perret
  - Centre Léon Bérard, Lyon
  - ICM Val d'Aurelle, Montpellier
  - ORACLE - Centre d'Oncologie de Gentilly, Nancy
  - Hôpital Privé du Confluent S.A.S., Nantes
  - Centre Antoine Lacassagne, Nice
  - Centre Hospitalier Régional d'Orléans, Orléans
  - Hôpital Saint-Louis, Paris
  - Hôpital Cochin, Paris
  - Institut du Cancer Courlancy Reims, Reims
  - Centre Eugène Marquis, Rennes
  - Centre Hospitalier de Saint-Brieuc, Saint-Brieuc
  - ICO Centre René Gauducheau, Saint-Herblain
  - Clinique Mutualiste de l'Estuaire, Cité Sanitaire, Saint-Nazaire
  - Institut de Cancérologie Lucien Neuwirth, Saint-Priest-en-Jarez
  - Hôpitaux Universitaires de Strasbourg, Strasbourg
  - ICL Institut de Cancérologie de Lorraine, Vandœuvre-lès-Nancy
  - Gustave Roussy, Villejuif

IPD SHARING:
Plan to Share IPD: No